CLINICAL TRIAL: NCT00057486
Title: A Pilot, Proof-of-Concept, Dose-Escalating Trial of Recombinant Human Interleukin-12 (rhIL-12) Versus Placebo Along With Paromomycin and Azithromycin for Chronic Cryptosporidiosis in AIDS
Brief Title: Interleukin 12 (IL-12) for the Treatment of Cryptosporidiosis in AIDS Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2R01AI041735-04A2 (NIH); 5R01AI041735-05 (NIH)
Record Dates: First submitted 2003-04-02; First posted 2003-04-03 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2003-03

CONDITIONS: HIV Infections; Cryptosporidiosis
Keywords: Chronic Diarrhea; Interleukin 12
MeSH Terms: conditions — HIV Infections; Cryptosporidiosis | interventions — Interleukin-12

INTERVENTIONS:
Drug: IL-12

SUMMARY:
There is no proven effective treatment for chronic diarrhea caused by the parasite Cryptosporidium in advanced AIDS. This trial will test the safety of interleukin-12 (IL-12) as part of a combination therapy for this parasite.

DETAILED DESCRIPTION:
Cryptosporidium parvum can cause chronic diarrhea and biliary disease in people with AIDS, resulting in significant morbidity and mortality. Highly effective antiparasitic treatment for this infection is not currently available. Paromomycin and azithromycin have some efficacy and have been used in combination in a small number of patients. However, in clinical trials of this drug combination, patients remained infected with the parasite despite improvement of their symptoms.

Improving the immune system with highly active antiretroviral therapy (HAART) has been the most effective therapy described for cryptosporidiosis (chronic infection with Cryptosporidium parvum), with over 80% of patients showing improvement. However, immune reconstitution is not possible in all patients.

Interferon gamma expression is strongly associated with control of cryptosporidiosis. IL-12 stimulates interferon gamma, and IL-12 treatment has been shown to prevent cryptosporidiosis in mice. This study will evaluate IL-12 in combination with standard therapy for cryptosporidiosis in patients with AIDS.

This is a dose-escalation study. All patients will be treated with paromomycin and azithromycin. The initial group will be treated with either 110 ng/kg IL-12 (6 patients) or placebo injections (2 patients) twice a week for 4 weeks. If the initial dose is ineffective and the combination of drugs is tolerated, a second group of patients will be randomized to either 300 ng/kg IL-12 (6 patients) or placebo injections (2 patients) twice a week for 4 weeks. Patients will be evaluated for eradication of the parasite (as measured by immunofluorescence and intestinal biopsy), decreases in stool frequency, decreases in 24 hour stool volume, stimulation of intestinal Th1 cytokine production, increases in body weight, improvements in Karnofsky score, and improvements in serum alkaline phosphatase levels and transaminases (if elevated at baseline).

ELIGIBILITY:
Inclusion criteria:

* HIV infection
* CD4 cell count < 150 cells/µl
* Stable antiretroviral regime that includes at least two nucleotide analogues for at least 4 weeks
* Viral load < 10,000 copies/ml
* Chronic diarrhea, defined as three loose or watery bowel movements a day for 5 days per week over 3 weeks
* Stool positive for Cryptosporidium and no other enteric pathogen (bacterial culture, C. difficile toxin assay, AFB stain, ova and parasite examination, and stain for microsporidia)
* Karnofsky score >= 70
* Acceptable methods of contraception

Exclusion Criteria:

* Pregnant
* Active opportunistic infection
* History of hypersensitivity or significant intolerance to aminoglycosides, macrolide antibiotics, or colony stimulating factors
* Requires intravenous fluids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2
Dates: Start 1997-09; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur White, Principal Investigator — Baylor College of Medicine